CLINICAL TRIAL: NCT04282421
Title: Survival in Patients Receiving Allogeneic Hematopoietic Stem Cell Transplantation for Myelofibrosis in Five French Centers
Brief Title: Survival in Myelofibrosis Patients After Allogeneic Hematopoietic Stem Cell Transplantation in Five Centers in France
Acronym: SYMFASCT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI014
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Myelofibrosis
Keywords: allogeneic hematopoietic stem cell transplantation; survival; graft versus host disease
MeSH Terms: conditions — Primary Myelofibrosis; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators would like to conduct a retrospective study in five centers in France in the goal to evaluate the survival of patients receiving allogeneic hematopoietic stem cell transplantation for myelofibrosis.

DETAILED DESCRIPTION:
The allogeneic stem cell transplantation is the only curative treatment for myelofibrosis. However, because of complications such as infection, graft-versus-host disease and conditioning toxicity, this procedure is associated with a high morbidity-mortality rate. The discovery of molecular and genetic markers permitted to improve therapeutic strategy and survival of patient in the last few years. In this study, the investigators want to make an overview of survival, incidence of relapse and incidence of acute and chronic graft versus host disease in allogeneic stem cell transplantation for myelofibrosis, in five centers in France, between 2007 and 2017.

ELIGIBILITY:
Inclusion Criteria: adult patients receiving allogeneic hematopoietic stem cell transplantation for myelofibrosis in five centers in France (Nancy, Besancon, Strasbourg, Pitie Salpetriere and Lyon) between 2007 and 2017

-

Exclusion Criteria:

* age < 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients receiving allogeneic hematopoietic stem cell transplantation for myelofibrosis in five centers in France (Nancy, Besançon, Strasbourg, Pitié Salpètrière and Lyon) between 2007 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
survival | at 1 year
  incidence of survival in the cohort

SECONDARY OUTCOMES:
incidence of relapse | at 1 year
  incidence of relapse in the cohort
incidence of acute graft versus host disease | at 3 months
  incidence of acute graft versus host disease in the cohort
incidence of chronic graft versus host disease | at 1 year
  incidence of chronic graft versus host disease in the cohort

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroger N, Panagiota V, Badbaran A, Zabelina T, Triviai I, Araujo Cruz MM, Shahswar R, Ayuk F, Gehlhaar M, Wolschke C, Bollin R, Walter C, Dugas M, Wiehlmann L, Lehmann U, Koenecke C, Chaturvedi A, Alchalby H, Stadler M, Eder M, Christopeit M, Gohring G, Koenigsmann M, Schlegelberger B, Kreipe HH, Ganser A, Stocking C, Fehse B, Thol F, Heuser M. Impact of Molecular Genetics on Outcome in Myelofibrosis Patients after Allogeneic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2017 Jul;23(7):1095-1101. doi: 10.1016/j.bbmt.2017.03.034. Epub 2017 Apr 4. PMID 28389256
- [Background] Hussein K, Stucki-Koch A, Alchalby H, Triviai I, Kroger N, Kreipe H. Cytokine Expression Pattern in Bone Marrow Microenvironment after Allogeneic Stem Cell Transplantation in Primary Myelofibrosis. Biol Blood Marrow Transplant. 2016 Apr;22(4):644-650. doi: 10.1016/j.bbmt.2015.12.006. Epub 2015 Dec 19. PMID 26708839